CLINICAL TRIAL: NCT06533150
Title: A Dopable Bioink for Augmented Tissue Engineering in Craniofacial Reconstruction, Innovative Pipeline for Drug Design and Selective Delivery Through Functionalized Polymeric Nanoparticles.
Brief Title: Functionalized Bioink Delivering Biomolecules for the Treatment of Craniofacial Diseases
Acronym: DART-CRAFT
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6830
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-07

CONDITIONS: Craniofacial Defects, Subtle; Skull Defect; Craniosynostoses
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient-derived cells isolated from tissue samples as well as tissue samples will be collected in biobanking infrastructures until the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: multiomic profiling — 2 aliquots of patients-derived bone tissue specimens (collected as surgical waste from routinely surgeries) will be collected and exploited from proteins and metabolites isolation according to standardized protocol. Then, samples will be digested using Filter-aided sample preparation digestion protocol and analysed by Liquid Chromatography Tandem Mass Spectrometry. Peptides will be loaded on the PepMap 100 C18 trap cartridge, and subsequently separated on an EASY Spray C18 analytical column. The mass spectrometer, equipped with a nanoESI spray source, operates in positive ion polarity and MS/MS mode. Also metabolites will be assessed by LC-MS/MS and will be separated by HPLC. Obtained results will be analyzed by integrated pathway analysis (IPA) to achieve the multiomic profiling of each patient thus identifying druggable targets to be exploited in drug design. The selected biomolecules will be then tested in patient cells using the developed bioink-nanoparticle complex.

SUMMARY:
The study aims to address the challenges of craniofacial bone reconstruction in pediatric and adult patients affected by congenital craniofacial malformations (i.e. craniosynostosis), trauma or tumors, by developing an innovative biohybrid material with tunable rheological properties, serving as a sealing agent and defect filler. Craniectomy/craniotomy procedures often leave bone defects that require cranioplasty to protect the underlying dura mater and the brain from physical insults. Reconstruction of the viscerocranial skeleton poses additional challanges, due to the complex anatomy of the facial skull and significant esthetic and functional demands on its reconstruction.

The study plans to develop a mouldable biosynthetic gelatin-methacrylamide (GelMA)-based hydrogel complexed with functionalized Poly (lactic-co-glycolic acid) (PLGA) nanoparticles for drug delivery. Osteoprogenitors cells (including mesenchymal stromal cells/osteoblasts and monocytes/osteoclasts) will be isolated from bone tissue fragments of enrolled patients and peripheral blood sample, respectively, to obtain 2D and 3D cultures mimicking the in vivo bone environment. High-throughput profiling of patients' samples will identify druggable targets for the bioactive compounds to be released by the bioink. In vitro validation will involve osteoprogenitor co-cultures derived from patients to assess uptake, release dynamics, biocompatibility, immunogenicity, and therapeutic effects of the developed complex. The final goal will be to develop a pre-prototype tissue engineering biocomposite for craniofacial bone reconstruction.

DETAILED DESCRIPTION:
To develop a mouldable biosynthetic collagen-based polymer matrix, commercial gelatin-methacrylamide (GelMA)-based hydrogels will be biochemically modified to finely tune their pseudo-plasticity and yield stress, and functionalized to implement drug delivery for improved biological properties. The GelMA will be chemically enriched with: adhesive molecules (e.g. alginate-based or ion releasing inorganic compounds), if needed, to increase the adhesion to implantable materials used in craniofacial reconstruction, thiol-based non- cleavage-type photoinitiators (e.g. eosinY combined with triethanolamine and vinyl caprolactam) to enable visible light-activated crosslinking and minimize the safety concerns of UV light. Photo-crosslinking will be achieved through a portable visible light device (420-480 nm) to induce the jellification of the bioink. The physical properties (morphology, viscoelastic properties, stiffness, resistance to an applied stress) of the different GelMA compounds will be analyzed according to standardized procedures. The adhesive properties of the GelMA will be measured by lap-shear strength tests in dry conditions. Once identified GelMA compounds showing the highest biological features, this will be endowed with functionalized Poly (lactic-co-glycolic acid) (PLGA)-based nanoparticles (NPs).

To this aim, biocompatible PLGA-Polyethylene glycol (PEG) NPs will be synthesized and functionalized with bis-sulfone for binding targeting moieties on the surface. The synthesis involves PLGA activation, PLGA-PEG conjugation, bis-sulfone activation, and PLGA-PEG-bis-sulfone conjugation. The PLGA/PEG ratio will be adjusted for the hydrophobicity/hydrophilicity payload. Bis-sulfone is used for selective and efficient PEGylation of protein's disulfide bond or to conjugate His-tagged protein/peptides according to standardized methods to implement either specific cell targeting or antimicrobial agents. High performance liquid chromatography (HPLC) will be used to validate the biosynthetic reaction. Dynamic Light Scattering (DLS), Nanoparticle Tracking Analysis (NTA), and Scanning electron microscopy (SEM) will define the morphological and ultrastructural properties of the final construct. Surface Plasmon Resonance will validate target recognition. Then, GelMA-NP hybrid compound assembly will be achieved through extrusion 3D printing according to standardized production pipelines. The hydrogel and the NP suspension will be dispensed through separate nozzles, in 2D and 3D patterns with 100-1000 nm feature sizes, under pressure and temperature control. Scalar NP concentrations will be used and then evaluated.

NP integrity and release dynamics of these from GelMA will be studied by submerging the GelMA-NPs loaded with fluorescent compound with a bio-mimetic cell growth medium and quantifying the NPs released in the supernatant in time course experiments. NP quantification will be performed using UV-Vis Spectroscopy, Fluorescence Spectroscopy or particle counting such as NTA system. NPs integrity will be studied with transmission electron microscopy (TEM) and DLS.

Once biochemically characterized GelMA-NPs, these will be used to deliver bioactive compounds identified through proteomics data as subsequently described.

To validate the developed bio-ink in in vitro craniofacial disease models, patients with craniofacial malformations undergoing cranial surgery will be selected and enrolled in the study. Specifically, paediatric patients affected by craniosynostosis and other inborn defects, trauma or brain tumors undergoing cranial surgery will be enrolled. Adult patients undergoing craniofacial surgery will be also selected and enrolled for craniofacial trauma and tumors. To this purpose, cranial bone tissue specimens derived from both paediatric and adult patients will be obtained as surgical waste during craniectomy or cranial vault remodeling upon obtaining the signed informed consent (by parents in case of children). For each patient, the waste tissues will be randomized into three aliquots. Of these, 1 aliquot will be collected in cell growth medium for seeding bone tissue samples into culture plate to isolate mesenchymal stromal cells (MSCs). Thereafter, MSC will be expanded up to the 3rd culture passage and collected in biobanking infrastructures with associated anonymized clinical data and optimized tracking system for subsequent analysis as follows. GelMA-based bioink NP release and biocompatibility will be analyzed using MSC, through functional assays to: evaluate focal adhesion dynamics and study cell adhesion to the gelified bioink by immunofluorescence assay. Cell behaviors and viability will be measured in time course experiments using a live cell imaging system (Incucyte Live Cells Analysis systems).

In addition, 2 aliquots of patients-derived bone tissue specimens will be snap-frozen in liquid nitrogen (after submerging it in cryoprotective medium with protease inhibitors). Proteins and metabolites will be isolated from these samples using in-house standardized protocol. Extracted samples will be then digested using Filter-aided sample preparation (FASP) digestion protocol. Then, samples will be analysed by Liquid Chromatography Tandem Mass Spectrometry (LC-MS/MS). Also metabolites will be assessed by LC-MS/MS and will be separated by HPLC. Then, obtained results on proteins and metabolites will be analysed by integrated pathway analysis (using IPA) to achieve the multiomic profiling of each patient thus identifying druggable targets to be exploited in drug design. Computational drug design tools, including molecular docking and virtual screening, will be employed to identify the lead compounds from drug/chemical databases capable of interacting with the selected targets from the integrated omic profile datasets. The dynamic behavior, stability, and binding interactions of target-ligand complexes will be studied through Molecular dynamics (MD) simulations to analyze binding motifs and hotspots. MD-informed insights on molecular interactions will guide the design and optimization of novel compounds. This will involve incorporating structural modifications with ligand-based approaches, and performing virtual screening to enhance binding affinity, selectivity, and drug-likeness. The biomolecules identified through these in silico studies will be then commercially purchased and encapsulated in PLGA NPs. In this regard, nanoprecipitation and single emulsion will be exploited for hydrophobic payloads, while double-emulsion solvent evaporation technique (w1/o/w2) will be employed for hydrophilic payloads. After, PLGA delivering selected compounds will be complexed into hydrogel (GelMA) matrix. The functional trophic and pro-regenerative properties of the bioink compound delivering biomolecules will be assessed in MSC to test osteogenic properties - through ALP activity assay, in vitro mineralization staining and marker gene expression analysis. In addition, human umbilical vein endothelial cells (commercial line) will be treated with GelMA-NPs-drug complex for evaluating the angiogenic properties by counting and sizing the capillary-like structures formed in vitro (tube formation assay).

In addition, a small aliquot of peripheral venous blood (2-3 ml for pediatric patients and up to 7 ml for adult patients) from routine clinical examinations will be collected. PBMCs will be isolated from whole blood sample using Ficoll density gradient centrifugation technique. Monocyte/macrophage cells will be then separated through CD14 antibody-conjugated magnetic beads and cultured in vitro with factors (i.e. M-CSF, RANKL) to form mature osteoclasts. These will be used to evaluate the bio-resorbability of GelMA-NP compound. Briefly, osteoclasts will be seeded on the GelMA-NP nanopatterned surfaces and the expression of typical osteoclast-specific markers will be assessed through immunofluorescence analysis. SEM and immunofluorescence assay will be used to visualize ultra-structurally the osteoclast-bioink interface and discriminate resorption two- and three-dimensionally.

MSC/osteoprogenitors and osteoclasts derived from patients will be also exploited to obtain 2D and 3D in vitro culture to mimic the biological microenviroment existing at the bone-implant boundary for the validation of the developed bioink complex. The bioink components will be either bioprinted with cells (i.e. cells delivered through an independent nozzle) to form cell-laden models, or printed on the growth surface of cell culture vessels and let jelify before cell seeding, according to the aims of each test. The release dynamics of NP from the GelMA, cell viability and proliferation, angiogenic and bone regenerative effects will be assessed as mentioned above.

To test its antibacterial effects, both the unloaded GelMA and the GelMA-NP will be printed on to petri dishes and let jelify. Thereafter it will be incubated with the opportunistic bacterial strains (E. coli, S. aureus, Streptococcus mutans, Enterococcus faecalis and Pseudomonas aeruginosa) in the appropriate culture broth overnight. Bacterial adhesion and count will be assessed comparatively, testing dose- and time-related effects. Antibacterial activity of GelMA-NP over GelMA, will be also supported by SEM imaging.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients (0-3 years) undergoing surgery for craniosynostosis and other inborn defects/trauma/brain tumors
* Adult patients (18-50 years) undergoing craniofacial surgery for (mainly) trauma and tumours

Exclusion Criteria:

* Paediatric patients older than 3 years of age
* Adults older than 50 years of age
* Paediatric patients and adult patients with other cranial diseases
* Patients with cranial defects that do not require craniofacial surgery

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients undergoing surgery for craniosynostosis and other inborn defects (e.g. trauma, brain tumors) as per standard of care. Adult patients affected by trauma and tumors undergoing craniectomy as per standard of care. Pediatic patient will be enrolled at Fondazione Policlinico Universitario A. Gemelli IRCCS and at Azienda Ospedaliera di Rilievo Nazionale (AORN) Santobono Pausilipon. Adult patient will be enrolled at Policlinico di Bari. Samples derived from180 patients will be analysed for this study, 60 patients per UO will be enrolled prospectively.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Development of bio-ink nanoparticles complex | 12 months
  Development of at least 50 gelatin-methacrylamide (GelMA)-based hydrogels bio-ink complexed with Poly (lactic-co-glycolic acid) (PLGA) nanoparticles (NPs) showing a sustained and prolonged NPs release from GelMA matrix for 15-20 days. The efficiency of the developed complex will be evaluated by submerging the GelMA-NPs loaded with fluorescent compound with a bio-mimetic cell growth medium and quantifying the NPs released in the surnatant in time course experiments. NP quantification will be performed using UV-Vis Spectroscopy, Fluorescence Spectroscopy or particle counting such as Nanoparticle Tracking Analysis (NTA). NPs integrity will be studied by transmission electron microscopy (TEM) and Dynamic Light Scattering (DLS).

SECONDARY OUTCOMES:
Development of bio-ink nanoparticles complex delivering selected biomolecules | 18 months
  Encapsulation/conjugation of a range from 5-10 biomolecules in at least 70% of PLGA nanoparticles incorporated within hydrogel matrix. The efficiency of the developed complex will be evaluated by submerging the GelMA-NPs loaded with biomolecules with a bio-mimetic cell growth medium and quantifying the NPs released in the surnatant in time course experiments. NP quantification will be performed using UV-Vis Spectroscopy, Fluorescence Spectroscopy or particle counting such as Nanoparticle Tracking Analysis (NTA). NPs integrity will be studied by transmission electron microscopy (TEM) and Dynamic Light Scattering (DLS).
Validation of the complex bio-ink efficiency in bone regeneration | 22 months
  Assessment of 90% cell viability and at least 2-fold increased levels of osteospecific marker expression and mineralized matrix deposition following in vitro treatments of cells with bio-ink-nanoparticle complexes in at least 20 of biological replicates compared to untreated cells (control). Cell viability will be measured by live/dead kit assay. The biological functionality of the complex consisting of GelMA-NPs-biomolecule(s) will be evaluated by gene expression analysis and bone matrix staining and its quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Massimi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC neurochirurgia Infantile, Roma, Italy